CLINICAL TRIAL: NCT00970151
Title: Determinants of Fetal Inflammatory Exposure at Term
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: March of Dimes (Other)
Responsible Party: Laura Goetzl, MD, Medical University of South Carolina
Other Study IDs: HR # 15251; 6-FY06-311
Record Dates: First submitted 2008-02-19; First posted 2009-09-02 (Estimated); Last update posted 2009-10-12 (Estimated); Status verified 2009-10

CONDITIONS: Maternal-Fetal Relations
Keywords: Fetal Inflammation; Birth Outcome; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, blood serum, placenta, spinal fluid (for some subjects)
Oversight: Data Monitoring Committee: No

SUMMARY:
The hypothesis of this study is that maternal and fetal biologic variation in the balance between pro-inflammatory and anti-inflammatory mediators can be measured by currently available techniques. In addition, the investigators hypothesize that a pro-inflammatory maternal phenotype increases the risk of fetal exposure to intrauterine hyperthemia and inflammatory cytokines; and that intrapartum events, especially known risk factors for fever at term such as epidural analgesia and prolonged rupture of membranes, may interact with underlying maternal factors to increase fetal exposure to inflammatory cytokines.

This experiment aims to establish the first large-scale cohort to evaluate biomarkers for maternal and fetal inflammation in term pregnancy and to elucidate the relative antepartum and intrapartum contributions to fetal inflammation.

DETAILED DESCRIPTION:
It has been demonstrated that intrapartum fever >100.4 degrees Fahrenheit is associated with increased maternal and fetal levels of interleukin-6 (IL-6) at delivery. Maternal and fetal IL-6 levels are highly correlated, and placental transport of cytokines has been demonstrated. While intrapartum fever is traditionally attributed to acquired infection (chorioamnionitis), our data indicate that the maternal inflammatory balance assessed prior to the onset of labor may be a significant determinant of subsequent intrapartum fever. The increased risk of neonatal brain injury may be cytokine mediated or may, in part, be secondary to increased vulnerability to hypoxic injury in the setting of elevated fetal brain temperature.

The baseline prevalence of intrapartum fever at term is 1-5%. Factors associated with an increased risk of intrapartum fever include maternal age, nulliparity (75%), Hispanic race, induction and longer labor. However, in recent years, the most potent risk factor for intrapartum fever has clearly been epidural analgesia - which is selected for intrapartum pain relief by the majority of mothers in the US especially in the first, most painful birth. We have demonstrated that the risk of fever after epidural analgesia increases with increasing duration of epidural analgesia - therefore, the risk of fever after epidural analgesia is largely confined to nulliparous women. Multiparous women deliver shortly after the onset of active labor, resulting in a short duration of exposure to epidural analgesia, and are not at increased risk. Randomized studies demonstrate that the independent contribution of epidural analgesia to intrapartum fever risk is 3 to 7-fold. Rates of intrapartum fever >100.4 degrees Fahrenheit in nulliparas with epidural analgesia range from 14.5% to 33%. Rates at the upper end of this range are observed in large, public hospitals with primarily Hispanic populations. Conversely, lower rates are observed at private hospitals with primarily Caucasian populations.

This study will make observations based upon:

1. 10 mL of blood drawn the day of enrollment
2. 10 mL of blood drawn upon admission to Labor and Delivery
3. A sample of spinal fluid if a spinal epidural is chosen by the patient
4. Blood collected from the placenta and umbilical cord

In addition, the mother's temperature will be taken every hour during labor.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparity
* Singleton gestation
* Full term (>37 weeks) pregnancy
* Vertex presentation
* Candidate for trial of labor
* Ability to provide informed consent

Exclusion Criteria:

* Multiple gestation
* Autoimmune Disease
* Treatment with anti-inflammatory agents during pregnancy

Ages: 14 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 600 racially and ethnically diverse nulliparas who present to the Prenatal Wellness Center at Cannon Place and Northwoods Clinic with a full term (>37 weeks) pregnancy and who deliver in the Labor and Delivery Suite at MUSC Hospital
Sampling Method: Probability Sample
Enrollment: 618 (Actual)
Dates: Start 2005-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Fetal exposure to inflammation as assessed by cord cytokine levels | During birth

CONTACTS AND LOCATIONS:
Overall Officials: Laura Goetzl, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical Univeristy of South Carolina, Charleston, South Carolina, United States